## Platelet-rich Plasma (PRP) for Endometrial Regeneration and Repair NCT02825849

Document Date: Nov 15, 2020

Summary of PRP Study Protocol

## Statistical Analysis Plan:

This study was a small, first-in-human pilot study of the use of Platelet Rich Plasma in women with either Asherman's syndrome or think uterine lining. Our over-arching goal was to establish the feasibility of administering and study the impact of PRP in a fertility clinic setting. The primary outcome of this study was improvements in uterine lining. Our secondary outcome was pregnancy rate. We ultimately enrolled 17 subjects into the intervention arm and 5 subjects into the control arm. This study was not powered to detect statistically significant differences. Accordingly, we have calculated and presented descriptive statistics of our baseline characteristics and study outomes. In particular, we have calculated means and standard deviation for continuous outcomes and percentages for dichotomous outcomes.